CLINICAL TRIAL: NCT01020864
Title: Phase II Trial of Cetuximab in Combination With Chemotherapy (Carboplatin and Navelbine) for Patients With Platinum-resistant Head and Neck Cancer
Brief Title: Cetuximab in Combination With Chemotherapy for Patients With Head and Neck Cancer
Acronym: CECAVI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.08
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Head and Neck Neoplasms
Keywords: Platinum-resistent head and neck cancer; Cetuximab; Carboplatin; Navelbine; Phase II trial; Combination chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Carboplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Patients will be treated with Cetuximab, Carboplatin and Vinorelbine i.v. day 1, every 2nd week.
  Patients will be treated until progression and/or in case of unacceptable toxicity or if the patient wishes to stop treatment.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: Vinorelbine

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 500 mg/m² i.v. day 1, every 2nd week
  Other Names: Erbitux
Drug: Carboplatin — Carboplatin AUC = 3 i.v. day 1, every 21nd week
Drug: Vinorelbine — Vinorelbine 25 mg/m² i.v. day 1, every 2nd week

SUMMARY:
This is an open, multicenter phase II study. The purpose is to demonstrate the efficacy of cetuximab in combination with carboplatin and vinorelbine as second line treatment in patients with recurrent or metastatic head and neck cancer who have progressed during or after treatment with first line cisplatinum.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified squamous cell carcinoma of the head and neck where curatively intended local treatment is not possible.
* Measurable or non-measurable disease.
* Disease progression during or after first line palliative chemotherapy with cisplatinum or patients with recurrence < 6 months after primary concomitant chemo-radiotherapy with cisplatinum.
* WHO Performance Status 0-2.
* Age ≥ 18 years.
* Neutrophil count (ANC) ≥ 1.5 x 10^9/l and platelets ≥ 100 x 10^9/l.
* Normal liver function with bilirubin < 1.5 x UNL (Upper Normal Limit), no UNL for ALAT with liver metastases.
* Creatinin clearance ≥ 50 ml/min.
* Signed informed consent.

Exclusion Criteria:

* Other active malignant disease.
* Patients who are considered unable to follow the treatment plan or follow-up visits.
* Other serious disease (e.g. severe heart disease, myocardial infarction (MI) within 1 year, active infection).
* Any condition or treatment which after the opinion of the investigator may expose the patient to a risk or may influence the purpose of the trial.
* Pregnant or lactating women.
* Known hypersensitivity towards one or more of the components of the treatment.
* Prior treatment with either cetuximab or other inhibitors of EGFR.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2.5 years
Response rate | 3 years

SECONDARY OUTCOMES:
Toxicity | 2.5 years
Median survival | 3 years
Correlation between response and evolvement in tumor biology markers. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, MD, PhD, Study Chair — Odense University Hospital
Locations (1):
- Department of Oncology, Odense University Hospital, Odense, Denmark